CLINICAL TRIAL: NCT06044909
Title: Multimodal Image Registration for Helping Laparoscopic Liver Surgery Guidance
Acronym: IMMORTALLS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN952023/CHUSTE
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Hepatectomy; Laparoscopy
Keywords: Intraoperative; preoperative; multimodal data; registration; laparoscopy; hepatectomy; augmented reality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing minimally invasive hepatectomy by conventional or robot-assisted laparoscopy: Patients undergoing minimally invasive hepatectomy by conventional or robot-assisted laparoscopy will be included.
  Interventions: Procedure: Minimal invasive hepatectomy, intraoperative stage; Procedure: Minimal invasive hepatectomy, postoperative stage; Other: Preoperative data collection; Other: Intraoperative data collection; Other: Postoperative data collection

INTERVENTIONS:
Procedure: Minimal invasive hepatectomy, intraoperative stage — Trocar layout is recorded by photo or diagram. The video of conventional or robot-assisted laparoscopy and intraoperative laparoscopic ultrasound images (where applicable) are recorded by the surgeon and anonymized. Depth measurements of internal structures (tumors, cysts, vascular network, anatomical landmarks) are taken using identifiable points on the surface of the liver for tumour resection.
Procedure: Minimal invasive hepatectomy, postoperative stage — The registration of imaging data in conventional or robot-assisted laparoscopy is performed by the scientific team using the developed registration algorithm. The data obtained from the clinical intervention will help improve the registration algorithm.
Other: Preoperative data collection — Patient code (anonymised) + inclusion number, repeated on each page. Anonymised CT or MRI scan and date of scan. Type of cancer, planned surgery and approach (robotic or laparoscopic). Patient's age. Patient's surgical history. Toxic habits: tobacco, alcohol. Healthy liver, liver disease, cirrhosis. Anticoagulant and antiaggregant treatment.
Other: Intraoperative data collection — Endoscope calibration. Intraoperative surgical and ultrasound images. Measurements for tumor's size and tumor's distances from liver surface and vascular vascular structures.
Other: Postoperative data collection — Definitive anatomical pathology with the measurement of resection margins.

SUMMARY:
Multimodal intraoperative minimal-invasive (laparoscopic or robotic) liver surgery images will be registered to each other. Explicitly, these are the ultrasound and laparoscope images. Once they are registered, they will reveal the hidden tumor's location to the surgeon in real time through augmented reality. The intraoperative augmentation will also be enriched with the preoperative data (e.g., CT or MRI). This will simplify minimal invasive liver surgery, improve surgical safety and accuracy. It will also shorten hospital stays and contribute to an overall better quality of life for the patient, which in return will reduce the health-care costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hepatectomy;
* Patients for whom good-quality imaging is available (CT scan and/or MRI and/or ultrasound);
* Patients over 18 years of age;
* Minimally invasive surgery by conventional or robot-assisted laparoscopy.

Exclusion Criteria:

* Surgery by laparotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing minimally invasive hepatectomy by conventional or robot-assisted laparoscopy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Analysis accuracy of the augmented reality by aligned with the intraoperative measurements | 28 months
  The accuracy of the augmented reality will be assessed based on how well the preoperative data will be aligned with the intraoperative measurements. In order to assess the accuracy, measurements of multiple distances between the center of mass (mean position) of different internal structures (tumors, anatomical vascular networks, anatomical landmarks) visible both in the preoperative imaging and in the intraoperative imaging will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand LE ROY, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No